CLINICAL TRIAL: NCT01545375
Title: Study to Determine Protective Efficacy Against Otitis Media and Assess Safety of an Investigational Pneumococcal Vaccine 2189242A in Healthy Infants
Brief Title: Evaluation of a Vaccine for Reducing Ear and Lung Infections in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115597; 2011-003956-38 (EudraCT Number)
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal
Keywords: nasopharyngeal carriage; safety; immunogenicity; US; Pneumococcal vaccine; efficacy; Streptococcus pneumoniae; infants
MeSH Terms: conditions — Streptococcal Infections | interventions — 13-valent pneumococcal vaccine; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dPly-PhtD Group (Experimental): Healthy Native American infants between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination, receiving GSK2189242A (dPly-PhtD) vaccine co-administered with Prevenar13™: 3 primary doses at 2, 4, 6 months of age and a booster dose at 12-15 months of age.
  PedvaxHIB was given as study vaccine to a subset of subjects at 2, 4 and 12-15 months.
  At the primary epoch, the dPly-PhtD vaccine was administered intramuscularly into the right anterolateral thigh and at the booster epoch, the dPly-PhtD vaccine was administered into the right deltoid or anterolateral thigh if the deltoid muscle size was not adequate.
  At the primary epoch, the co-administered Prevenar13™ and PedvaxHIB vaccines were administered intramuscularly into the left anterolateral thigh and at the booster epoch, the Prevenar13™ and PedvaxHIB vaccines were administered into the left deltoid or anterolateral thigh if the deltoid muscle size was not adequate.
  Interventions: Biological: Pneumococcal vaccine GSK2189242A; Biological: Prevnar 13®; Biological: PedvaxHIB®
- Control Group (Placebo Comparator): Healthy Native American infants between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination, receiving Placebo vaccine co-administered with Prevenar13™: 3 primary doses at 2, 4, 6 months of age and a booster dose at 12-15 months of age.
  PedvaxHIB was given as study vaccine to a subset of subjects at 2, 4 and 12-15 months.
  At the primary epoch, the Placebo vaccine was administered intramuscularly into the right anterolateral thigh and at the booster epoch, the Placebo vaccine was administered into the right deltoid or anterolateral thigh if the deltoid muscle size was not adequate.
  At the primary epoch, the co-administered Prevenar13™ and PedvaxHIB vaccines were administered intramuscularly into the left anterolateral thigh and at the booster epoch, the Prevenar13™ and PedvaxHIB vaccines were administered into the left deltoid or anterolateral thigh if the deltoid muscle size was not adequate.
  Interventions: Biological: Placebo; Biological: Prevnar 13®; Biological: PedvaxHIB®

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2189242A — 4 doses administered intramuscularly
  Arms: dPly-PhtD Group
Biological: Placebo — 4 doses administered intramuscularly
  Arms: Control Group
Biological: Prevnar 13® — 4 doses administered intramuscularly
Biological: PedvaxHIB® — 4 doses administered intramuscularly

SUMMARY:
The purpose of this study is to 1) demonstrate the protective efficacy against acute otitis media (AOM), 2) assess safety of the GlaxoSmithKline (GSK) Biologicals' pneumococcal vaccine GSK2189242A in Native American infants aged less than 24 months, living in the southwestern US, in and around the Navajo and White Mountain Apache reservations, and 3) evaluate the impact on acute lower respiratory tract infections (ALRI) up to the second year of life.

DETAILED DESCRIPTION:
The study will also evaluate the impact of the pneumococcal vaccine GSK2189242A on nasopharyngeal carriage in a subgroup of children called Carriage subgroup. Immunogenicity and reactogenicity of the pneumococcal vaccine GSK2189242A will be evaluated in another subgroup of children called Immuno/reacto subgroup.

Protocol Posting has been updated following Protocol Amendment 3, April 2012, leading to the addition of a secondary outcome measure.

Protocol Posting has been updated following Protocol Amendment 7, March 2017, to add serological testing for antibodies against the Hib polysaccharide PRP on samples collected 12 months following booster dose (Month 22) in the Immuno/reacto sub-cohort, in order to evaluate the long term persistence of immune responses to co-administered PedvaxHIB vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject who the investigator believes that their parent(s)/Legally Authorized Representative(s) (LARs) can and will comply with the requirements of the protocol.
* A male or female American Indian infant between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Voluntary, written informed consent obtained from the parents/LAR(s) of the subject. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by a witness.
* Healthy subject as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of more than 35 6/7 weeks.

Exclusion Criteria:

For all infants:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol starting from 30 days before each dose and ending 30 days after each dose of study vaccines, with the exception of licensed inactivated influenza vaccines and recommended pediatric vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against S. pneumoniae.
* Obstruction or anomalies of the nasopharyngeal space.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s) including latex.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Any medical or social condition which might interfere with the assessment of the study objectives in the opinion of the investigator.

For infants in the Immuno/reacto subgroup only:

• Previous vaccination against H. influenzae type b.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1806 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Chinle, Arizona
  - GSK Investigational Site, Fort Defiance, Arizona
  - GSK Investigational Site, Whiteriver, Arizona
  - GSK Investigational Site, Gallup, New Mexico
  - GSK Investigational Site, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammitt LL, Campbell JC, Borys D, Weatherholtz RC, Reid R, Goklish N, Moulton LH, Traskine M, Song Y, Swinnen K, Santosham M, O'Brien KL. Efficacy, safety and immunogenicity of a pneumococcal protein-based vaccine co-administered with 13-valent pneumococcal conjugate vaccine against acute otitis media in young children: A phase IIb randomized study. Vaccine. 2019 Dec 3;37(51):7482-7492. doi: 10.1016/j.vaccine.2019.09.076. Epub 2019 Oct 16. PMID 31629570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1806 subjects were enrolled in this study, Three sub-cohorts of subjects were foreseen: Immuno/reacto sub-cohort for assessment of immunogenicity, Carriage sub-cohort for assessment of impact on carriage of S. pneumoniae and "No additional procedures" sub-cohort comprising subjects not included in any of the above sub-cohorts.
Pre-assignment Details: Out of the 1806 subjects enrolled in this study, 1803 were vaccinated and therefore included in the Total Vaccinated Cohort. 3 subjects were excluded for the following reasons: one subject had an invalid Inform Consent form and 2 subjects received subject number but did not receive any vaccine dose.
Period: Overall Study
Arm/Group | dPly-PhtD Group | Control Group
Started | 900 | 903
Completed | 803 | 813
Not Completed | 97 | 90
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 34 | 31
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 58 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dPly-PhtD Group | Control Group | Total
Number analyzed (Participants) | 900 | 903 | 1803
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.7 (1.69) | 7.6 (1.65) | 7.6 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 459 | 441 | 900
  Male | 441 | 462 | 903
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American indian or Alaskan native: American Indian or Alaskan Native | 900 | 903 | 1803

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Any Acute Otitis Media (AOM) Diagnosed and Verified Against American Academic of Pediatrics (AAP) Criteria
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/sum of follow-up expressed in years (T[year)]). Definition of clinical AOM diagnosed and verified against AAP criteria required meeting three criteria based on the guidelines from the AAP [AAP, 2004], as per the judgment of a treating physician or equivalent licensed medical professional: A history of acute (recent, usually abrupt) onset of signs and symptoms of middle-ear inflammation and middle-ear effusion (MEE).AND The presence of MEE indicated by any of the following: a) Bulging of tympanic membrane; b) Limited or absent mobility of tympanic membrane; c) Air-fluid level behind tympanic membrane; d) Otorrhea AND Signs or symptoms of middle-ear inflammation as indicated by either: a) Distinct erythema of tympanic membrane or b) Distinct otalgia (discomfort clearly referable to the ear[s] that resulted in interference with or precluded normal activity or sleep).
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: Analysis was performed on the modified according to protocol cohort for efficacy which included all evaluable subjects for whom data concerning efficacy outcome measures were available (efficacy cohort) and for whom non-compliance with the vaccination intervals during primary vaccination was the only elimination criterion from the efficacy cohort.
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.425 | 0.442
Statistical Analysis 1: Comparison: dPly-PhtD Group vs Control Group; VE-AOM against AAP criteria: Occurrence of AOM during efficacy follow-up period was compared between groups to estimate Vaccine Efficacy (VE) and its 95% confidence interval using the Anderson & Gill model (generalization of Cox proportional hazard model) taking into account for recurrent events [Kelly, 2000]. VE= (1 - hazard ratio) x 100 Censoring occurred at the time of the last scheduled or medically attended visit; Test type: Superiority — The objective was to demonstrate that VE induced by GSK2189242A vaccine (three doses in the first year of life and a booster dose in the second year of life)in preventing clinical AOM diagnosed and verified against AAP criteria was greater than 0%, as compared to the control group. One-sided p-value for the Wald-Test obtained from the general Cox proportional hazard model was calculated; p = 0.3016, Regression, Cox — The primary objective was met if the one-sided p-value calculated for the null hypothesis H0=[clinical AOM VE ≤ 0%] was lower than defined 1-sided alpha level: (17.8%); Vaccine Efficacy = 3.81, 95% CI 2-sided [-11.35 to 16.90]

2. Secondary Outcome: Time to Occurrence of Any Episodes of AOM Diagnosed by Healthcare-provider
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/sum of follow-up expressed in years (T[year)]). A healthcare-provider-diagnosed clinical AOM case was defined as an AOM event diagnosed by a treating physician or equivalent licensed medical professional with or without clinical symptoms documented in the routine medical record.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: Analysis was performed on the modified ATP cohort for efficacy which included all evaluable subjects for whom data concerning efficacy outcome measures were available (efficacy cohort) and for whom non-compliance with the vaccination intervals during primary vaccination was the only elimination criterion from the efficacy cohort.
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.678 | 0.699

3. Secondary Outcome: Time to Occurrence of Any Clinical Acute Otitis Media (AOM) Diagnosed and Verified Against Modified American Academic of Pediatrics (AAP) Criteria
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/sum of follow-up expressed in years (T[year)]). Definition of clinical AOM diagnosed and verified against modified AAP criteria required a history of acute disease (i.e. AAP criterion 1) together with abnormal tympanic membrane (i.e. one of the AAP criteria 2 or 3a), as per the judgment of a treating physician or equivalent licensed medical professional: 1. A history of acute (recent, usually abrupt) onset of signs and symptoms of middle-ear inflammation and middle-ear effusion (MEE).AND 2. The presence of MEE that is indicated by any of the following: a) Bulging of tympanic membrane, b) Limited or absent mobility of tympanic membrane, c) Air-fluid level behind tympanic membrane, d) Otorrhea OR 3. Signs or symptoms of middle-ear inflammation as indicated by: a) Distinct erythema of tympanic membrane.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: as for outcome 2
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.567 | 0.599

4. Secondary Outcome: Number of Subjects With Any Recurrent Healthcare Provider Diagnosed Acute Otitis Media (AOM)
Description: Recurrent AOM was defined as at least 3 AOM episodes diagnosed by a physician or equivalent licensed medical professional and occurring within 6 months or at least 4 episodes within one year, regardless of the etiology.
Time Frame: From the administration of dose 1 up to Month 22
Population: Analysis was performed on the Total vaccinated cohort which included all subjects who had received at least one vaccination dose.
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 900 | 903
Participants | 30 | 32

5. Secondary Outcome: Time to Occurrence of Any Draining Acute Otitis Media (AOM)
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/sum of follow-up expressed in years (T[year)]). Draining AOM was defined as AOM with otorrhea or with spontaneously perforated tympanic membrane. In this case, middle ear fluid (MEF) was to be swabbed with no tympanocentesis needed and tested for the presence of S. pneumoniae and other pathogens as part of the routine clinical practice. Draining pneumococcal AOM were defined as draining AOM cases with S. pneumoniae identified in MEF.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: Analysis was performed on the modified ATP for efficacy which included all evaluable subjects for whom data concerning efficacy outcome measures were available (efficacy cohort) and for whom non-compliance with the vaccination intervals during primary vaccination was the only elimination criterion from the efficacy cohort.
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.055 | 0.060

6. Secondary Outcome: Time to Occurrence of Any Draining Pneumococcal Acute Otitis Media (AOM)
Description: as for outcome 5
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: as for outcome 5
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.008 | 0.006

7. Secondary Outcome: Number of Subjects With Any Acute Otitis Media (AOM) With Temporally Related Carriage
Description: AOM with temporally related carriage was defined as AOM with nasopharyngeal swab taken within 3 days before or after an AOM episode.
Time Frame: From the administration of dose 1 up to Month 22
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 900 | 903
Participants | 338 | 368

8. Secondary Outcome: Time to Occurrence of Medically Attended Acute Lower Respiratory Tract Infection (ALRI)
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/ sum of follow-up expressed in years (T[year)]). ALRI was defined by the presence of tachypnea (respiratory rate >50 amongst children 2 to 12 months of age, and respiratory rate >40 in children over 1 year of age) and at least two of the following signs and symptoms: cough; fever documented at visit or reported within preceding 3 days (Fever was defined as temperature ≥100.4°F (38.0°C) regardless of the route of measurement); increased work of breathing: grunting, nasal flaring, and intercostal and/or subcostal retractions; auscultatory abnormalities: wheezing, crackles, rhonchi, decreased breath sounds.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: as for outcome 2
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.143 | 0.141

9. Secondary Outcome: Time to Occurrence of Medically Attended ALRI With Fever Documented at the Visit or History of Fever Within 3 Days Preceding a Given Episode
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/ sum of follow-up expressed in years (T[year)]). ALRI was defined by the presence of tachypnea (respiratory rate >50 amongst children 2 to 12 months of age, and respiratory rate >40 in children over 1 year of age) and at least two of the following signs and symptoms: cough; fever documented at visit or reported within preceding 3 days (Fever is defined as temperature ≥100.4°F (38.0°C) regardless of the route of measurement); increased work of breathing: grunting, nasal flaring, and intercostal and/or subcostal retractions; auscultatory abnormalities: wheezing, crackles, rhonchi, decreased breath sounds.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: as for outcome 2
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.109 | 0.105

10. Secondary Outcome: Time to Occurrence of Any Medically Attended Healthcare-provider-diagnosed ALRI With Fever Documented at the Visit or History of Fever Within 3 Days Preceding a Given Episode.
Description: Time to occurrence of any episode of AOM is expressed in terms of rate: Person-year rate = number of episodes (n)/ sum of follow-up expressed in years (T[year)]). A healthcare-provider-diagnosed ALRI with fever case was defined as, but not limited to, chest infection, bronchiolitis, pneumonia, bronchopneumonia, pleural effusion or empyema diagnosed by a treating physician or equivalent licensed medical professional with fever documented at the time of visit or history of fever within 3 days preceding a given episode and with or without other clinical symptoms documented in the routine medical record.
Time Frame: Any time from 2 weeks after the administration of dose 3 up to Month 22
Population: as for outcome 2
Measure: Number; unit: Episodes per person-year
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 808 | 831
Episodes per person-year | 0.253 | 0.259

11. Secondary Outcome: Number of Subjects With S. Pneumoniae (Any and Serotype Specific) in the Nasopharynx - Carriage Sub-cohort
Description: Positive cultures of S. pneumoniae (any and serotype specific) identified in the nasopharynx were analyzed.
Time Frame: At 7 months of age (Month 5), 12-15 months of age (Month 10),18-22 months of age (Month 16) and 24-27 months of age (Month 22)
Population: Analysis was performed on the Total vaccinated cohort for carriage which included around 400 subjects not included in the immuno/reacto sub-cohort, who had received at least one vaccination dose and for whom data concerning carriage outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 355 | 359
Participants
  Month 5 | 202 | 224
  Month 10: number analyzed (Participants) | 349 | 353
  Month 10 | 201 | 213
  Month 16: number analyzed (Participants) | 343 | 342
  Month 16 | 192 | 213
  Month 22: number analyzed (Participants) | 336 | 346
  Month 22 | 204 | 223

12. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (Ply) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - Immuno/Reacto Sub-cohort
Description: Anti-Ply and anti-PhtD antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA) immunoassay and expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). Cut-off of the assay were concentrations equal to (=) 12 EL.U/mL for anti-Ply antibodies and = 17 EL.U/mL for anti-PhtD antibodies.
Time Frame: One month post-dose 3 [PIII(Month 5)], prior to booster dose [PIII(Month 10)] and one and twelve months post-booster dose [Post-booster(Month 11) and Post-booster(Month 22)], respectively
Population: Analysis was performed on the ATP cohort for immunogenicity which included all evaluable subjects from the Immuno/reacto sub-cohort (composed of 200 subjects from each study group) for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 116 | 120
EL.U/mL
  Anti-Ply-PIII (Month 5) | 24206.23 [21618.31 to 27103.95] | 1063.15 [853.29 to 1324.63]
  Anti-Ply-Pre-booster (Month 10): number analyzed (Participants) | 115 | 114
  Anti-Ply-Pre-booster (Month 10) | 13108.68 [10959.48 to 15679.36] | 2245.92 [1845.51 to 2733.21]
  Anti-Ply-Post-booster (Month 11): number analyzed (Participants) | 115 | 115
  Anti-Ply-Post-booster (Month 11) | 36234.97 [33306.01 to 39421.51] | 2658.05 [2191.75 to 3223.55]
  Anti-Ply-Post-booster (Month 22): number analyzed (Participants) | 114 | 117
  Anti-Ply-Post-booster (Month 22) | 19390.01 [17011.67 to 22100.85] | 4639.15 [3954.54 to 5442.29]
  Anti-PhtD-PIII (Month 5) | 4144.62 [3469.43 to 4951.20] | 989.65 [778.36 to 1258.29]
  Anti-PhtD-Pre-booster (Month 10): number analyzed (Participants) | 115 | 114
  Anti-PhtD-Pre-booster (Month 10) | 2625.77 [2189.20 to 3149.41] | 2271.53 [1730.59 to 2981.55]
  Anti-PhtD-Post-booster (Month 11): number analyzed (Participants) | 115 | 115
  Anti-PhtD-Post-booster (Month 11) | 8680.76 [7489.85 to 10061.04] | 2324.28 [1768.42 to 3054.87]
  Anti-PhtD-Post-booster (Month 22): number analyzed (Participants) | 114 | 117
  Anti-PhtD-Post-booster (Month 22) | 5248.38 [4650.71 to 5922.86] | 5535.93 [4776.89 to 6415.59]

13. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid (Ply) Haemolysis Activity, or Hem-Ply Antibodies
Description: Inhibition of Ply hemolysis activity was not evaluated due to assay stability issues.
Time Frame: as for outcome 12
Population: The analysis was to be performed on the according to protocol cohort for immunogenicity. But inhibition of Ply hemolysis activity was not evaluated due to assay stability issues.
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl Ribitol Phosphate (Anti-PRP) - Immuno/Reacto Sub-cohort
Description: Seroprotection rate = Anti-PRP antibody concentrations ≥ 0.15 µg/mL.
Time Frame: 1 month post-dose 3 [PIII(Month 5)], prior to booster dose [PIII(Month 10)], 1 month post-booster dose [Post-booster(Month 11)], 12 months post-booster dose [Post-booster(Month 22)]
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 115 | 119
µg/mL
  Anti-PRP PIII (Month 5): number analyzed (Participants) | 114 | 119
  Anti-PRP PIII (Month 5) | 4.65 [3.40 to 6.34] | 6.66 [5.02 to 8.85]
  Anti-PRP Pre-booster (Month 10): number analyzed (Participants) | 115 | 114
  Anti-PRP Pre-booster (Month 10) | 0.90 [0.69 to 1.19] | 1.12 [0.85 to 1.46]
  Anti-PRP Post-booster (Month 11): number analyzed (Participants) | 103 | 104
  Anti-PRP Post-booster (Month 11) | 12.32 [9.02 to 16.82] | 17.28 [13.15 to 22.69]
  Anti-PRP Post-booster (Month 22): number analyzed (Participants) | 113 | 115
  Anti-PRP Post-booster (Month 22) | 1.51 [1.16 to 1.95] | 1.84 [1.48 to 2.29]

15. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F
Description: Antibody concentrations were measured by Electro-chemiluminescence assay (ECL), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was a serotype-specific antibody concentration higher than or equal to (≥) LLOQ (Lower Limit of Quantification) expressed in µg/mL: 0.08 for Anti-1; 0.075 for anti-3; 0.061 for Anti-4; 0.198 for Anti-5; 0.111 for Anti-6A and Anti-18C; 0.102 for Anti-6B; 0.063 for Anti-7F; 0.066 for Anti-9V; 0.160 for Anti-14; 0.199 for Anti-19A; 0.163 for Anti-19F; 0.073 for Anti-23F.
Time Frame: One month post-dose 3 [PIII(Month 5)], prior to booster dose [PIII(Month 10)] and one month post-booster dose [Post-booster(Month 11)]
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 112 | 118
µg/mL
  Anti-1 PIII(Month 5) | 3.35 [2.91 to 3.86] | 3.18 [2.8 to 3.62]
  Anti-1 Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-1 Pre-Booster (Month 10) | 0.57 [0.5 to 0.65] | 0.55 [0.49 to 0.62]
  Anti-1 Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-1 Post-Booster (Month 11) | 4.45 [3.83 to 5.17] | 4.83 [4.16 to 5.59]
  Anti-3 PIII(Month 5): number analyzed (Participants) | 111 | 118
  Anti-3 PIII(Month 5) | 0.59 [0.52 to 0.67] | 0.52 [0.47 to 0.58]
  Anti-3 Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-3 Pre-Booster (Month 10) | 0.16 [0.14 to 0.20] | 0.13 [0.11 to 0.15]
  Anti-3 Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-3 Post-Booster (Month 11) | 0.66 [0.59 to 0.75] | 0.57 [0.51 to 0.64]
  Anti-4 PIII(Month 5) | 2.05 [1.79 to 2.35] | 1.98 [1.75 to 2.24]
  Anti-4 Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-4 Pre-Booster (Month 10) | 0.34 [0.3 to 0.38] | 0.31 [0.27 to 0.35]
  Anti-4 Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-4 Post-Booster (Month 11) | 3.98 [3.35 to 4.73] | 3.85 [3.23 to 4.59]
  Anti-5 PIII(Month 5): number analyzed (Participants) | 106 | 115
  Anti-5 PIII(Month 5) | 2.4 [2.09 to 2.77] | 2.41 [2.12 to 2.73]
  Anti-5 Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-5 Pre-Booster (Month 10) | 0.66 [0.58 to 0.76] | 0.61 [0.53 to 0.69]
  Anti-5 Post-Booster (Month 11): number analyzed (Participants) | 106 | 106
  Anti-5 Post-Booster (Month 11) | 4.24 [3.68 to 4.89] | 3.98 [3.48 to 4.56]
  Anti-6A PIII(Month 5) | 5.27 [4.55 to 6.11] | 4.74 [4.13 to 5.43]
  Anti-6A Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-6A Pre-Booster (Month 10) | 0.97 [0.85 to 1.11] | 0.9 [0.78 to 1.03]
  Anti-6A Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-6A Post-Booster (Month 11) | 10.31 [9.0 to 11.82] | 10.28 [8.89 to 11.89]
  Anti-6B PIII(Month 5) | 3.5 [2.9 to 4.23] | 3.31 [2.74 to 4.0]
  Anti-6B Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-6B Pre-Booster (Month 10) | 0.66 [0.56 to 0.79] | 0.64 [0.54 to 0.76]
  Anti-6B Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-6B Post-Booster (Month 11) | 10.03 [8.68 to 11.6] | 9.62 [8.24 to 11.25]
  Anti-7F PIII(Month 5) | 4.47 [3.99 to 5.0] | 4.35 [3.87 to 4.89]
  Anti-7F Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-7F Pre-Booster (Month 10) | 0.89 [0.79 to 1.01] | 0.87 [0.78 to 0.97]
  Anti-7F Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-7F Post-Booster (Month 11) | 6.61 [5.81 to 7.53] | 6.65 [5.82 to 7.59]
  Anti-9V PIII(Month 5) | 2.22 [1.89 to 2.62] | 2.24 [1.97 to 2.53]
  Anti-9V Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-9V Pre-Booster (Month 10) | 0.43 [0.37 to 0.5] | 0.45 [0.39 to 0.52]
  Anti-9V Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-9V Post-Booster (Month 11) | 4.14 [3.52 to 4.88] | 4.38 [3.78 to 5.08]
  Anti-14 PIII(Month 5) | 8.46 [7.04 to 10.16] | 8.78 [7.67 to 10.04]
  Anti-14 Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-14 Pre-Booster (Month 10) | 1.79 [1.51 to 2.11] | 1.83 [1.6 to 2.1]
  Anti-14 Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-14 Post-Booster (Month 11) | 13.22 [11.35 to 15.4] | 13.14 [11.22 to 15.39]
  Anti-18C PIII(Month 5) | 2.51 [2.20 to 2.87] | 2.33 [2.05 to 2.64]
  Anti-18C Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-18C Pre-Booster (Month 10) | 0.38 [0.33 to 0.44] | 0.34 [0.29 to 0.39]
  Anti-18C Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-18C Post-Booster (Month 11) | 5.41 [4.63 to 6.32] | 5.28 [4.46 to 6.25]
  Anti-19A PIII(Month 5): number analyzed (Participants) | 111 | 117
  Anti-19A PIII(Month 5) | 2.65 [2.29 to 3.06] | 2.86 [2.46 to 3.33]
  Anti-19A Pre-Booster (Month 10): number analyzed (Participants) | 108 | 110
  Anti-19A Pre-Booster (Month 10) | 0.57 [0.47 to 0.68] | 0.61 [0.5 to 0.74]
  Anti-19A Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-19A Post-Booster (Month 11) | 7.64 [6.58 to 8.87] | 8.07 [6.92 to 9.42]
  Anti-19F PIII(Month 5) | 3.61 [3.18 to 4.09] | 3.60 [3.17 to 4.09]
  Anti-19F Pre-Booster (Month 10): number analyzed (Participants) | 112 | 111
  Anti-19F Pre-Booster (Month 10) | 0.78 [0.67 to 0.92] | 0.84 [0.72 to 0.98]
  Anti-19F Post-Booster (Month 11): number analyzed (Participants) | 112 | 111
  Anti-19F Post-Booster (Month 11) | 7.96 [6.92 to 9.17] | 8.23 [7.13 to 9.49]
  Anti-23F PIII(Month 5): number analyzed (Participants) | 110 | 116
  Anti-23F PIII(Month 5) | 1.97 [1.64 to 2.36] | 2.04 [1.72 to 2.43]
  Anti-23F Pre-Booster (Month 10): number analyzed (Participants) | 109 | 108
  Anti-23F Pre-Booster (Month 10) | 0.36 [0.3 to 0.43] | 0.39 [0.32 to 0.47]
  Anti-23F Post-Booster (Month 11): number analyzed (Participants) | 109 | 108
  Anti-23F Post-Booster (Month 11) | 3.71 [3.16 to 4.36] | 3.97 [3.27 to 4.83]

16. Secondary Outcome: Antibody Concentrations Against Vaccine-related Serotypes 6C
Description: No analysis was performed on antibody concentrations against vaccine-related serotype 6C as no specific qualified/validated assay was available.
Time Frame: as for outcome 15
Population: The analysis was to be performed on the ATP cohort for immunogenicity. But no analysis was performed for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay was available.
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) LLOQ: 8 for OPA-1, OPA-3 and OPA-6B; 33 for OPA-4, and OPA-14; 50 for OPA-5; 151 for OPA-6A; 330 for OPA-7F; 275 for OPA-9V; 11 for OPA-18C; 143 for OPA-19A; 36 for OPA-19F; 101 for OPA-23F.
Time Frame: One month post-dose 3 [PIII(Month 5)] and one month post-booster dose [Post-booster(Month 11)]
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 57 | 59
Titers
  OPA-1 PIII(Month 5): number analyzed (Participants) | 49 | 57
  OPA-1 PIII(Month 5) | 76.0 [43.0 to 134.4] | 32.9 [20.2 to 53.7]
  OPA-1 Post-Booster (Month 11): number analyzed (Participants) | 56 | 48
  OPA-1 Post-Booster (Month 11) | 191.0 [114.9 to 317.7] | 219.7 [134.7 to 358.5]
  OPA-3 PIII(Month 5): number analyzed (Participants) | 41 | 52
  OPA-3 PIII(Month 5) | 319.9 [233.3 to 438.8] | 190.1 [140.9 to 256.7]
  OPA-3 Post-Booster (Month 11): number analyzed (Participants) | 39 | 39
  OPA-3 Post-Booster (Month 11) | 452.4 [342.1 to 598.3] | 399.5 [294.1 to 542.5]
  OPA-4 PIII(Month 5): number analyzed (Participants) | 55 | 58
  OPA-4 PIII(Month 5) | 1450.4 [1159.2 to 1814.7] | 1397.8 [1136.3 to 1719.3]
  OPA-4 Post-Booster (Month 11): number analyzed (Participants) | 55 | 49
  OPA-4 Post-Booster (Month 11) | 2657.2 [2254.7 to 3131.6] | 2592.5 [2167.7 to 3100.5]
  OPA-5 PIII(Month 5): number analyzed (Participants) | 47 | 54
  OPA-5 PIII(Month 5) | 792.7 [610.0 to 1030.0] | 464.7 [337.7 to 639.4]
  OPA-5 Post-Booster (Month 11): number analyzed (Participants) | 53 | 49
  OPA-5 Post-Booster (Month 11) | 1541.5 [1254.2 to 1894.8] | 1192.6 [857.8 to 1658.0]
  OPA-6A PIII(Month 5): number analyzed (Participants) | 52 | 57
  OPA-6A PIII(Month 5) | 4945.3 [3877.7 to 6306.7] | 5231.7 [4349.7 to 6292.6]
  OPA-6A Post-Booster (Month 11): number analyzed (Participants) | 49 | 46
  OPA-6A Post-Booster (Month 11) | 9149.5 [7640.0 to 10957.2] | 10266.5 [8902.8 to 11839.1]
  OPA-6B PIII(Month 5): number analyzed (Participants) | 55 | 59
  OPA-6B PIII(Month 5) | 2754.9 [2168.1 to 3500.4] | 2140.1 [1443.9 to 3172.1]
  OPA-6B Post-Booster (Month 11): number analyzed (Participants) | 56 | 49
  OPA-6B Post-Booster (Month 11) | 5909.9 [4895.5 to 7134.4] | 5663.3 [4502.2 to 7123.9]
  OPA-7F PIII(Month 5): number analyzed (Participants) | 46 | 57
  OPA-7F PIII(Month 5) | 8429.3 [6931.1 to 10251.3] | 7539.0 [6295.3 to 9028.4]
  OPA-7F Post-Booster (Month 11): number analyzed (Participants) | 36 | 33
  OPA-7F Post-Booster (Month 11) | 10746.6 [9081.4 to 12717.2] | 9504.8 [7707.8 to 11720.7]
  OPA-9V PIII(Month 5): number analyzed (Participants) | 51 | 54
  OPA-9V PIII(Month 5) | 2391.3 [1699.5 to 3364.6] | 2728.4 [2002.2 to 3718.1]
  OPA-9V Post-Booster (Month 11): number analyzed (Participants) | 50 | 45
  OPA-9V Post-Booster (Month 11) | 6001.1 [4904.8 to 7342.4] | 6206.9 [4806.4 to 8015.5]
  OPA-14 PIII(Month 5): number analyzed (Participants) | 53 | 59
  OPA-14 PIII(Month 5) | 2236.4 [1722.1 to 2904.2] | 1988.5 [1437.7 to 2750.3]
  OPA-14 Post-Booster (Month 11): number analyzed (Participants) | 57 | 50
  OPA-14 Post-Booster (Month 11) | 3981.9 [3233.2 to 4904.0] | 3856.0 [3011.3 to 4937.7]
  OPA-18C PIII(Month 5): number analyzed (Participants) | 52 | 58
  OPA-18C PIII(Month 5) | 1927.9 [1532.7 to 2425.1] | 1736.2 [1346.8 to 2238.1]
  OPA-18C Post-Booster (Month 11): number analyzed (Participants) | 52 | 48
  OPA-18C Post-Booster (Month 11) | 4240.3 [3345.8 to 5374.0] | 4349.6 [3437.7 to 5503.4]
  OPA-19A PIII(Month 5): number analyzed (Participants) | 48 | 57
  OPA-19A PIII(Month 5) | 2204.4 [1626.0 to 2988.4] | 2060.2 [1590.9 to 2668.0]
  OPA-19A Post-Booster (Month 11): number analyzed (Participants) | 48 | 46
  OPA-19A Post-Booster (Month 11) | 5630.3 [4474.1 to 7085.2] | 6447.5 [5235.0 to 7941.0]
  OPA-19F PIII(Month 5): number analyzed (Participants) | 52 | 58
  OPA-19F PIII(Month 5) | 1355.0 [1018.9 to 1802.1] | 1112.4 [785.0 to 1576.2]
  OPA-19F Post-Booster (Month 11): number analyzed (Participants) | 54 | 48
  OPA-19F Post-Booster (Month 11) | 3222.8 [2513.5 to 4132.2] | 2574.0 [1838.8 to 3603.2]
  OPA-23F PIII(Month 5): number analyzed (Participants) | 52 | 58
  OPA-23F PIII(Month 5) | 3072.8 [2473.1 to 3817.9] | 2634.9 [1991.9 to 3485.5]
  OPA-23F Post-Booster (Month 11): number analyzed (Participants) | 52 | 50
  OPA-23F Post-Booster (Month 11) | 6240.2 [5555.3 to 7009.4] | 5958.6 [5117.3 to 6938.2]

18. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 6C
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine-related pneumococcal serotypes 6C (OPA-6C). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 145.
Time Frame: One month post-dose 3 [PIII(Month 5)] and one month post-booster dose [Post-booster(Month 11)]
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 45 | 54
Titers
  OPA-6C PIII(Month 5) | 3161.8 [2369.0 to 4219.8] | 2616.6 [1924.2 to 3558.2]
  OPA-6C Post-Booster (Month 11): number analyzed (Participants) | 38 | 38
  OPA-6C Post-Booster (Month 11) | 5151.0 [4003.5 to 6627.3] | 5637.2 [4436.4 to 7163.1]

19. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, After Primary Vaccination - Immuno/Reacto Sub-cohort
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). The Immuno /reacto sub-cohort was composed of 200 vaccinated subjects from each study group.
Time Frame: Within the 4-day (Days 0-3) post-primary vaccination period following each dose
Population: Analysis was performed on Immuno/reacto sub-cohort which included around 200 subjects from the total vaccinated cohort, for whom at least one vaccination dose was documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 198 | 197
Participants
  Any Pain, post Dose 1 | 149 | 131
  Grade 3 Pain, post Dose 1 | 38 | 36
  Any Redness, post Dose 1 | 59 | 58
  Grade 3 Redness, post Dose 1 | 0 | 0
  Any Swelling, post Dose 1 | 35 | 28
  Grade 3 Swelling, post Dose 1 | 0 | 0
  Any Pain, post Dose 2: number analyzed (Participants) | 181 | 185
  Any Pain, post Dose 2 | 137 | 139
  Grade 3 Pain, post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Pain, post Dose 2 | 29 | 43
  Any Redness, post Dose 2: number analyzed (Participants) | 181 | 185
  Any Redness, post Dose 2 | 54 | 63
  Grade 3 Redness, post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Redness, post Dose 2 | 0 | 0
  Any Swelling, post Dose 2: number analyzed (Participants) | 181 | 185
  Any Swelling, post Dose 2 | 48 | 34
  Grade 3 Swelling, post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Swelling, post Dose 2 | 0 | 0
  Any Pain, post Dose 3: number analyzed (Participants) | 172 | 171
  Any Pain, post Dose 3 | 96 | 96
  Grade 3 Pain, post Dose 3: number analyzed (Participants) | 172 | 171
  Grade 3 Pain, post Dose 3 | 12 | 20
  Any Redness, post Dose 3: number analyzed (Participants) | 172 | 171
  Any Redness, post Dose 3 | 61 | 51
  Grade 3 Redness, post Dose 3: number analyzed (Participants) | 172 | 171
  Grade 3 Redness, post Dose 3 | 1 | 0
  Any Swelling, post Dose 3: number analyzed (Participants) | 172 | 171
  Any Swelling, post Dose 3 | 42 | 27
  Grade 3 Swelling, post Dose 3: number analyzed (Participants) | 172 | 171
  Grade 3 Swelling, post Dose 3 | 1 | 0

20. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, After Booster Vaccination - Immuno/Reacto Sub-cohort
Description: as for outcome 19
Time Frame: Within the 4-day (Days 0-3) post-booster vaccination period
Population: Analysis was performed on Immuno/reacto sub-cohort which included around 200 subjects from the total vaccinated cohort, for whom the booster vaccination dose was documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 156 | 153
Participants
  Any Pain | 100 | 83
  Grade 3 Pain | 24 | 18
  Any Redness | 59 | 60
  Grade 3 Redness | 0 | 0
  Any Swelling | 39 | 37
  Grade 3 Swelling | 0 | 0

21. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination, After Primary Vaccination - Immuno/Reacto Sub-cohort
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness (Irr./Fuss.), Loss of appetite (Loss Appet.) and Fever (axillary route - temperature equal or higher than [≥] 38.0 degrees Celsius [°C]),. Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = (axillary) temperature higher than (>) 40.0°C. Related = Occurrence of the specified symptom assessed by the investigator as causally related to vaccination. The Immuno /reacto sub-cohort was composed of 200 vaccinated subjects from each study group.
Time Frame: Within the 4-day (Days 0-3) post-primary vaccination period following each dose
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 198 | 197
Participants
  Any Drowsiness, post Dose 1 | 97 | 94
  Grade 3 Drowsiness, post Dose 1 | 12 | 8
  Related Drowsiness, post Dose 1 | 91 | 91
  Any Irr./Fuss., post Dose 1 | 129 | 122
  Grade 3 Irr./Fuss., post Dose 1 | 13 | 17
  Related Irr./Fuss., post Dose 1 | 123 | 115
  Any Loss Appet., post Dose 1 | 46 | 42
  Grade 3 Loss Appet., post Dose 1 | 3 | 3
  Related Loss Appet., post Dose 1 | 44 | 40
  Any Fever, post Dose 1 | 15 | 18
  Grade 3 Fever, post Dose 1 | 0 | 0
  Related Fever, post Dose 1 | 10 | 10
  Any Drowsiness, post Dose 2: number analyzed (Participants) | 181 | 185
  Any Drowsiness, post Dose 2 | 87 | 94
  Grade 3 Drowsiness, post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Drowsiness, post Dose 2 | 11 | 3
  Related Drowsiness, post Dose 2: number analyzed (Participants) | 181 | 185
  Related Drowsiness, post Dose 2 | 81 | 90
  Any Irr./Fuss., post Dose 2: number analyzed (Participants) | 181 | 185
  Any Irr./Fuss., post Dose 2 | 125 | 127
  Grade 3 Irr./Fuss., post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Irr./Fuss., post Dose 2 | 19 | 25
  Related Irr./Fuss., post Dose 2: number analyzed (Participants) | 181 | 185
  Related Irr./Fuss., post Dose 2 | 117 | 117
  Any Loss Appet., post Dose 2: number analyzed (Participants) | 181 | 185
  Any Loss Appet., post Dose 2 | 46 | 50
  Grade 3 Loss Appet., post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Loss Appet., post Dose 2 | 1 | 4
  Related Loss Appet., post Dose 2: number analyzed (Participants) | 181 | 185
  Related Loss Appet., post Dose 2 | 43 | 46
  Any Fever, post Dose 2: number analyzed (Participants) | 181 | 185
  Any Fever, post Dose 2 | 17 | 23
  Grade 3 Fever, post Dose 2: number analyzed (Participants) | 181 | 185
  Grade 3 Fever, post Dose 2 | 0 | 1
  Related Fever, post Dose 2: number analyzed (Participants) | 181 | 185
  Related Fever, post Dose 2 | 14 | 14
  Any Drowsiness, post Dose 3: number analyzed (Participants) | 172 | 172
  Any Drowsiness, post Dose 3 | 64 | 72
  Grade 3 Drowsiness, post Dose 3: number analyzed (Participants) | 172 | 172
  Grade 3 Drowsiness, post Dose 3 | 13 | 8
  Related Drowsiness, post Dose 3: number analyzed (Participants) | 172 | 172
  Related Drowsiness, post Dose 3 | 60 | 66
  Any Irr./Fuss., post Dose 3: number analyzed (Participants) | 172 | 172
  Any Irr./Fuss., post Dose 3 | 101 | 96
  Grade 3 Irr./Fuss., post Dose 3: number analyzed (Participants) | 172 | 172
  Grade 3 Irr./Fuss., post Dose 3 | 20 | 18
  Related Irr./Fuss., post Dose 3: number analyzed (Participants) | 172 | 172
  Related Irr./Fuss., post Dose 3 | 91 | 87
  Any Loss Appet., post Dose 3: number analyzed (Participants) | 172 | 172
  Any Loss Appet., post Dose 3 | 45 | 39
  Grade 3 Loss Appet., post Dose 3: number analyzed (Participants) | 172 | 172
  Grade 3 Loss Appet., post Dose 3 | 10 | 3
  Related Loss Appet., post Dose 3: number analyzed (Participants) | 172 | 172
  Related Loss Appet., post Dose 3 | 40 | 36
  Any Fever, post Dose 3: number analyzed (Participants) | 172 | 172
  Any Fever, post Dose 3 | 10 | 18
  Grade 3 Fever, post Dose 3: number analyzed (Participants) | 172 | 172
  Grade 3 Fever, post Dose 3 | 0 | 0
  Related Fever, post Dose 3: number analyzed (Participants) | 172 | 172
  Related Fever, post Dose 3 | 8 | 11

22. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination, After Booster Vaccination - Immuno/Reacto Sub-cohort
Description: as for outcome 21
Time Frame: Within the 4-day (Days 0-3) post-booster vaccination period
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 156 | 154
Participants
  Any Drowsiness | 65 | 65
  Grade 3 Drowsiness | 13 | 12
  Related Drowsiness | 60 | 56
  Any Irr./Fuss. | 97 | 86
  Grade 3 Irr./Fuss. | 27 | 16
  Related Irr./Fuss. | 89 | 74
  Any Loss Appet. | 43 | 41
  Grade 3 Loss Appet. | 6 | 7
  Related Loss Appet. | 41 | 30
  Any Fever | 8 | 15
  Grade 3 Fever | 0 | 0
  Related Fever | 7 | 9

23. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) After Primary Vaccination - Immuno/Reacto Sub-cohort
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination. The Immuno/reacto sub-cohort was composed of 200 vaccinated subjects from each study group.
Time Frame: Within the 31-day (Days 0-30) period post primary vaccination, across doses
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 200 | 200
Participants | 114 | 114

24. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) After Booster Vaccination - Immuno/Reacto Sub-cohort
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination. The Immuno /reacto sub-cohort was composed of 200 vaccinated subjects from each study group.
Time Frame: Within the 31-day (Days 0-30) period post booster vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 178 | 174
Participants | 53 | 47

25. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: An SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization, as per the medical or scientific judgement of the physician. Any = Occurrence of an SAE, regardless of relationship to vaccination.
Time Frame: From Day 0 to Month 22
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | dPly-PhtD Group | Control Group
Number analyzed (Participants) | 900 | 903
Participants | 229 | 232

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within the 4-day (Days 0-3) post-vaccination period; Unsolicited AEs: within the 31-day (Days 0-30) post-vaccination period; SAEs: during the whole study period (from Day 0 to Month 22).
Groups:
- dPly/PhtD Group: Healthy Native American infants between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination, receiving GSK2189242A (dPly-PhtD) vaccine co-administered with Prevenar13™: 3 primary doses at 2, 4, 6 months of age and a booster dose at 12-15 months of age. PedvaxHIB was given as study vaccine to a subset of subjects at 2, 4 and 12-15 months. At the primary epoch, the dPly-PhtD vaccine was administered intramuscularly into the right anterolateral thigh and at the booster epoch, the dPly-PhtD vaccine was administered into the right deltoid or anterolateral thigh if the deltoid muscle size was not adequate. At the primary epoch, the co-administered Prevenar13™ and PedvaxHIB vaccines were administered intramuscularly into the left anterolateral thigh and at the booster epoch, the Prevenar13™ and PedvaxHIB vaccines were administered into the left deltoid or anterolateral thigh if the deltoid muscle size was not adequate.
Arm/Group | dPly/PhtD Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/900 | 0/903
Serious Adverse Events (participants affected / at risk) | 229/900 | 232/903
Other Adverse Events (participants affected / at risk) | 191/200 | 189/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dPly/PhtD Group (N=900) | Control Group (N=903)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Benign familial neonatal convulsions (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sandifer's syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Developmental delay (General disorders) | 0 (0) | 1 (1)
Fever neonatal (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 3 (3)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 76 (97) | 74 (88)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4) | 6 (7)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 17 (17) | 17 (17)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 11 (11) | 12 (12)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 16 (17) | 13 (13)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 74 (87) | 53 (66)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 5 (5)
Pneumonia viral (Infections and infestations) | 4 (4) | 3 (3)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (4) | 5 (5)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 50 (51) | 67 (69)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (4)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Blood culture positive (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 13 (13)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clear cell sarcoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 14 (18) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 6 (6) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (9)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dPly/PhtD Group (N=200) | Control Group (N=200)
Conjunctivitis (Infections and infestations) | 12 (13) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 103 (180) | 98 (172)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 11 (12) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 12 (13) | 7 (8)
Erythema (Skin and subcutaneous tissue disorders) | 103 (235) | 109 (233)
Irritability (Psychiatric disorders) | 169 (458) | 166 (436)
Pain (General disorders) | 179 (482) | 175 (450)
Pyrexia (General disorders) | 87 (141) | 98 (170)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 10 (12)
Somnolence (Nervous system disorders) | 135 (313) | 146 (325)
Swelling (General disorders) | 88 (164) | 81 (126)
Teething (Gastrointestinal disorders) | 12 (15) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 59 (74) | 50 (58)
Viral infection (Infections and infestations) | 22 (26) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.